CLINICAL TRIAL: NCT07100665
Title: Effects of Intravenous Lidocaine Treatment on Sleep and Quality of Life in Fibromyalgia: An Observational Study
Acronym: pain
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Fibromyalgia, sleep quality
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Lidocaine Infusion; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Effects of Intravenous Lidocaine Treatment on Sleep and Quality of Life in Fibromyalgia:

SUMMARY:
Fibromyalgia (FM) is a psychosocial disorder characterized by widespread body pain, sleep disturbances, morning stiffness, and fatigue, impairing patients' quality of life. It is more common in middle-aged women, but its prevalence is 2% in the general population. Genetic factors, peripheral and central sensitization, autonomic nervous system dysfunction, and hypothalamic-pituitary axis dysregulation are thought to play important roles in its pathophysiology. In FM patients, decreased levels of norepinephrine, dopamine, serotonin, and some other neurotransmitters in the central nervous system and cerebrospinal fluid have been observed .

Complaints in FM patients vary considerably. The pain often begins localized and progresses to widespread body pain. Physical examination frequently reveals allodynia and hyperalgesia. Irritable bowel syndrome, depression, primary headaches, restless leg syndrome, Reynoud phenomenon, dry mouth, palpitations, allergic conditions, sexual dysfunction, dysmenorrhea, chronic fatigue syndrome, and anxiety disorder may accompany the condition. While these diagnoses are also considered in the differential diagnosis, their presence does not exclude the diagnosis of FM. The 2016 revised American College of Rheumatology (ACR) criteria are frequently used for diagnosis.

A multimodal approach is applied to treatment. These approaches include lifestyle changes, exercise, meditation, balneotherapy, yoga, psychotherapies, medical, and interventional methods. Antidepressants are often preferred for medical treatment. Patients' noncompliance with medication and side effects contribute to medical treatment failure. Acupuncture, dry needling, trigger point injections, and some complementary medicine methods are interventional methods .

In recent years, particularly in chronic pain management, intravenous (IV) methods are thought to reduce both peripheral and central sensitization. Intravenous drug therapies for chronic pain have been reported to be beneficial in addition to medical and interventional treatments. Magnesium, lidocaine, and ketamine are frequently administered IV treatments. There are various recommendations regarding the frequency and dosage of these medications, but a consensus has not yet emerged. IV lidocaine has been used in FM patients in recent years, although the number of studies reported is limited .

The symptom severity and pain prevalence in FM patients vary from patient to patient. Therefore, the treatment approach should be individualized. Sleep and quality of life disturbances frequently accompany FM and exacerbate other symptoms .

To our knowledge, IV lidocaine treatment is considered beneficial in FM patients, but we have not found any studies in the literature on its effectiveness on sleep and quality of life. In this study, we aimed to present the effects of IV lidocaine, a less frequently administered but well-established treatment method in FM, a challenging disease.

DETAILED DESCRIPTION:
In this study, after obtaining approval from the clinical research ethics committee (Health Sciences University Istanbul Kanuni Sultan Süleyman Training and Research Hospital, KAEK/2024.10.212), 51 patients aged 18-65 years who were treated with IV lidocaine and met the ACR (American College of Rheumatology) 2016 FM diagnostic criteria with accompanying sleep disturbance (Pittsburgh Sleep Quality Index score >5) and persistent complaints despite pharmacological and non-pharmacological FM treatments (Numeric Rating Scala >4) were retrospectively evaluated between June 2023 and June 2024 .. The study was conducted in accordance with the Declaration of Helsinki. Written informed consent was obtained from all patients in the study, which was conducted in a tertiary pain clinic in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guideline. Patient information was recorded: age, gender, body mass index, duration of symptoms, antineuropathic medical treatments, side effects observed during treatment, and pre- and post-treatment scores from the Fibromyalgia Impact Questionnaire (FIQ) at 4 and 12 weeks, the NRS-11 (Numeric Rating Scale), the Short Form-12 (SF-12) subcomponents of the Mental Component Scale-12 (MBS-12) and Physical Component Scale-12 (FBS-12), and the Pittsburgh Sleep Quality Index (PSQI).

Procedure The patient was taken to the procedure room, monitored (5-lead electrocardiogram (ECG), pulse oximetry, and blood pressure), and intravenous access was established in the forearm. Before IV lidocaine was administered, a 12-lead ECG was obtained and evaluated for dysrhythmia by a cardiologist with at least 10 years of experience. The patients were informed about possible side effects such as dizziness, vertigo, nausea and vomiting, numbness of the tongue, palpitations, a metallic taste in the mouth, and dry mouth. Patients were administered a 120-minute IV lidocaine infusion with 500 cc of 0.9% saline solution under appropriate monitoring conditions. Patients were monitored for 2 hours after the infusion. Patients received 5 mg/kg IV lidocaine twice weekly, 3 days apart, in accordance with current literature. The patients' FIQ, NRS-11, SF-12, and PSQI scores were recorded before and after treatment, 4 and 12 weeks.

Assessment Scales The FIQ is a 10-item scale ranging from 0 to 100, with each question rated on a 0 to 10 scale. Higher scores indicate increased disease activity (11). The NRS-11 is an 11-point numerical scale that allows patients to rate their pain on a scale from 0 (no pain at all) to 10 (the most severe pain they have ever experienced) .

The SF-12 consists of 12 questions: two questions on physical role, two on physical functioning, one on bodily pain, one on general health, one on energy, one on social functioning, two on emotional role, and two on mental health. The subcomponents of the SF-12, the FQI-12 and MQI-12, both have scores ranging from 0 to 100, with higher scores representing better health .

The PSQI is an index in which patients self-report their sleep quality and disturbances over a 1-month period. This index, consisting of 19 questions and 7 subheadings, is scored on a scale of 0-21, with 0 being the best and 3 being the worst. Higher scores indicate worse sleep quality and disturbances .

ELIGIBILITY:
Inclusion Criteria:Patients with sleep disturbances (Pittsburgh Sleep Quality Index score >5),

* who continued to have complaints despite pharmacological and non-pharmacological treatments for FM (Numeric Rating Scale >4),
* who met the ACR (American College of Rheumatology) 2016 FM diagnostic criteria,
* and who received IV lidocaine treatment,

Exclusion Criteria:-Patients whose medical treatment was changed during follow-up related to FM, those with metabolic diseases (chronic renal and hepatic failure, spondyloarthropathies, uncontrolled diabetes and hypertension, hypo/hyperthyroidism, etc.),

* patients with abnormal serum electrolyte levels, those taking magnesium or vitamin D supplements, pregnant women,
* patients with known allergy to the administered drug, those with malignancy or active infection, patients with neuromuscular disease and psychosis,
* patients with known cardiac arrhythmia and decompensated heart disease, -patients whose IV lidocaine treatment could not be completed,
* patients whose data were not available and who did not accept treatment were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty-two patients aged 18-65 years who were treated with IV lidocaine and met the ACR (American College of Rheumatology) 2016 FM diagnostic criteria and had ongoing complaints despite pharmacological and non-pharmacological FM treatments (Numeric Rating Scale >5) and accompanied by sleep disturbance (Pittsburgh Sleep Quality Index score >5) between June 2023 and June 2024 were evaluated retrospectively.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
NRS-11 (Numeric Rating Scale):It is an 11-point numerical scale on which patients can rate their pain from 0 (no pain at all) to 10 (the most severe pain they have ever felt). | 3 months

SECONDARY OUTCOMES:
Fibromyalgia impact questionnaire (FIQ) | 3 months
  The FIQ is a 10-item scale with scores ranging from 0 to 100, with each question rated on a scale of 0 to 10. A higher score indicates increased disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: halil ibrahim altun, specialist, Principal Investigator — Kanuni Sultan Süleyman Training and Research Hospital
Locations (1):
- İKanuni Sultan Süleyman Training and Research Hospital, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided